CLINICAL TRIAL: NCT04249102
Title: Prospective Randomized Clinical Study Assessing the Clinical Impact of Continuous vs Flash Glucose Monitoring During a 8 Weeks Period in Children, Adolescents and Young Adults 4 to 20 Years Old With Type 1 Diabetes Previously Using Flash Glucose Monitoring
Brief Title: Prospective Randomized Clinical Trial Assessing the Short Term Clinical Impact of Continuous vs Flash Glucose Monitoring in Children, Adolescents and Young Adults With Type 1 Diabetes
Acronym: GluMoCAY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CGM2020/1
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio either in the control group (Flash Glucose Monitoring system) or in the investigational group (Continuous Glucose Monitoring system).
  Randomization will be stratified according to the subject impaired hypoglycaemia awareness score (< 4 vs ≥ 4)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM Group (Experimental): The study group will be provided with a Continuous Glucose Monitoring system (Guardian Connect from Medtronic).
  Interventions: Device: Guardian Connect, Medtronic
- FGM Group (Active Comparator): The control group will be provided with a Flash Glucose Monitoring system (Abbott Diabetes Care).
  Interventions: Device: Abbott Diabetes Care

INTERVENTIONS:
Device: Guardian Connect, Medtronic — Guardian Connect is real-time continuous glucose sensor systems which provide glucose information updated every 5 minutes
  Arms: CGM Group
Device: Abbott Diabetes Care — Abbott Diabetes Care is a Flash Glucose Monitoring system that provides up to 8 hours of retrospective continuous glucose monitoring data to users when the monitor is waved in proximity with the sensor.
  Arms: FGM Group

SUMMARY:
Impaired hypoglycemia awareness, a significant problem for children with type 1 diabetes, is defined as neurogenic symptom response before autonomic response to hypoglycemia. Avoiding hypoglycemia appears to restore hypoglycemia awareness.

Investigators have previously demonstrated in a retrospective study that Flash Glucose Monitoring system decreased the risk of severe hypoglycemia in type 1 diabetic children and adolescents, even though Flash Glucose Monitoring system, unlike Continuous Glucose Monitoring system, does not provide glucose alerts.

Continuous Glucose Monitoring system, by providing real-time data with alarms, could benefit to subjects still experiencing severe hypoglycemia with Flash Glucose Monitoring system. Besides, in adults, Continuous Glucose Monitoring system reduced more effectively impaired hypoglycemia awareness compared to Flash Glucose Monitoring system.

In that context, investigators would like to assess the impact of Continuous Glucose Monitoring system instead of Flash Glucose Monitoring system on hypoglycemia in children and adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
All subjects will start with a 7 days run-in phase using their current Flash Glucose Monitoring System associated with a blind Continuous Glucose Monitoring system (Envision, Medtronic).

After one week, subjects randomized in the the interventional group will be provided with the Continuous Glucose Monitoring (Guardian Connect, Medtronic) and trained by dedicated diabetes educators for Continuous Glucose Monitoring usage including insertion of the sensor, calibration of the device twice daily and interpretation of the data. Subjects will use the sensors according to the license.

For both groups, insulin doses decisions are made by the participant according the received education.

After one week, all subjects will be contacted by phone focusing on the use of the technology. The treatment period is 8 weeks. The last week of the treatment period, subjects will use the blind Continuous Glucose Monitoring system (Envision, Medtronic) in addition to their allocated Glucose Monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged from 4 to 20 years
* Subjects with onset of diabetes before 16 years of age
* Diabetes duration of more than 1 year
* Subject currently using Flash Glucose Monitoring system in daily practice

Exclusion Criteria:

* Subject with mental disability
* Previous use of Continuous Glucose Monitoring system
* Subject currently participating to another clinical study

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the change in baseline hypoglycemia after 8-week Continuous Glucose Monitoring system use | At Baseline and after 8 weeks of Continuous Glucose Monitoring system use
  % of Time-Below-Range (i.e. < 70 mg/dl)

SECONDARY OUTCOMES:
To evaluate the change in severe hypoglycemia frequency in patients using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  Number of severe hypoglycaemia (i.e. hypoglycemic event leading leading to loss of consciousness)
To evaluate the change in HbA1c in patients monitored with Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  HbA1c value in %
To evaluate the change in glycemic variability in patients monitored with Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  % of time spent in the target range (70 - 180 mg/dl)
To evaluate the change in glycemic variability in patients monitored with Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  % of time spent above the target range (> 180 mg/dl and > 250 mg/dl)
To evaluate the change in glycemic variability in patients monitored with Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  % of time spent below the target range (< 70 mg/dl and < 54 mg/dl)
To evaluate the change in glycemic variability in patients monitored with Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  Coefficient of variation (SD/Mean)
To evaluate the change in glycemic variability in patients monitored with Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  low blood glucose index
To evaluate the change in the quality of life of patients using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  EQ-5D-3L Questionnaire
To evaluate the change in severe hypoglycemia frequency in patients with and without impaired hypoglycemia awareness using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  Number of severe hypoglycaemia (i.e. hypoglycemic event leading leading to loss of consciousness)
To evaluate the change in HbA1c in patients with and without impaired hypoglycemia awareness using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  HbA1c value in %
To assess the change in glycemic variability in patients with and without impaired hypoglycemia awareness using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  % of time spent in the target range (70 - 180 mg/dl)
To assess the change in glycemic variability in patients with and without impaired hypoglycemia awareness using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  % of time spent above the target range (> 180 mg/dl and > 250 mg/dl)
To assess the change in glycemic variability in patients with and without impaired hypoglycemia awareness using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  % of time spent below the target range (< 70 mg/dl and < 54 mg/dl)
To assess the change in glycemic variability in patients with and without impaired hypoglycemia awareness using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  Coefficient of variation (SD/Mean)
To assess the change in glycemic variability in patients with and without impaired hypoglycemia awareness using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  low blood glucose index
To evaluate the change in the quality of life of patients with and without impaired hypoglycemia awareness using Continuous Glucose Monitoring system in comparison to Flash Glucose Monitoring system. | At baseline and after 8 weeks of Continuous Glucose Monitoring system use
  EQ-5D-3L Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anissa Messaaoui, MD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Messaaoui A, Tenoutasse S, Hajselova L, Crenier L. Comparison Between Continuous Versus Flash Glucose Monitoring in Children, Adolescents, and Young Adults with Type 1 Diabetes: An 8-Week Prospective Randomized Trial. Diabetes Ther. 2022 Sep;13(9):1671-1681. doi: 10.1007/s13300-022-01297-x. Epub 2022 Jul 23. PMID 35870074